CLINICAL TRIAL: NCT00725907
Title: Treatment of ATFL Tears After Ankle Sprains With PRP
Brief Title: Treatment of ATFL Tears With PRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: "Meir" Medical Center, Kfar Saba, Israel, "Meir" Medical Center, Kfar Saba, Israel
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 6000; MeirMc07om0091CTIL
Record Dates: First submitted 2008-07-29; First posted 2008-07-31 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-07

CONDITIONS: Soft Tissue Healing
Keywords: PRP; ATFL

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- 1 (Experimental): PGRF
  Interventions: Biological: PGRF
- 2 (Placebo Comparator): saline
  Interventions: Biological: placebo saline

INTERVENTIONS:
Biological: PGRF — injection of 6cc into injured area
  Arms: 1
Biological: placebo saline — injection of 6cc into injured area
  Arms: 2

SUMMARY:
PRP will enhance ATFL tears healing by time and quality.

ELIGIBILITY:
Inclusion Criteria:

* athletes 18-30 years old 1st sprain within 3 days from injury

Exclusion Criteria:

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
time to return to active sport | 2

CONTACTS AND LOCATIONS:
Overall Officials: omer mei-dan, MD, Study Director — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel